CLINICAL TRIAL: NCT02180074
Title: Measurement of Distinct Biological Pools of Hydrogen Sulfide in Women With Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Christopher Kevil, Professor, Louisiana State University Health Sciences Center Shreveport
Other Study IDs: SRKH2SPOOLS
Record Dates: First submitted 2014-03-18; First posted 2014-07-02 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2014-06

CONDITIONS: Cardiovascular Disease
Keywords: Hydrogen Sulfide Pools,
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma.

GROUPS / COHORTS (5):
- I: Women without PAD (ABI >1.0 and <1.4) or CAD, and < 2 risk factors for cardiovascular disease (to serve as healthy controls)
- II: Women without PAD (ABI>1.0 and <1.4) or CAD and > 2 risk factors for cardiovascular disease
- III: Women with PAD as defined by ABI <0.9 and a coronary angiogram without any significant coronary artery disease.
- IV: Women with CAD without PAD, as defined by >50% stenosis by coronary angiography and ABI >1.0 and <1.4.
- V: Women with both CAD and PAD.

SUMMARY:
Cardiovascular disease which includes coronary artery disease and peripheral artery disease remains the leading cause of death among women in the United States. The impact of cardiovascular in women was not recognized by clinicians for a long time. It is now evident that, women suffer the consequences of cardiovascular at rates at least as high as those observed in men but there are still major gaps in our understanding this disease in women. Hydrogen sulfide (H2S), a gaseous mediator plays an important role in the cardiovascular system. Research has demonstrated it's critical role in animal ischemia reperfusion models. Hydrogen sulfide exists in distinct biological pools in blood. Recently, the Kevil lab has pioneered the development of new analytical techniques for accurate measurement of all biological pools of H2S. By measuring these distinct pools of H2S in women with and without cardiovascular disease the investigators hope to further understanding of role of H2S in pathophysiology of cardiovascular disease. This research will help to assess the ability of H2S and its distinct biological pools to potentially be a diagnostic marker or a therapeutic target for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting to the cardiac catheterization laboratory for coronary or peripheral angiography.
2. Females,Age>40years

Exclusion Criteria:

1. Inability to provide informed consent.
2. STelevationmyocardialinfarction.
3. Cardiogenicshock.

3. ABI >1.4 (indicative of non-compressible vessel needing further evaluation to diagnose PAD), unless documented known PAD. 4. Non-atheroscleroticPAD(e.g.Buerger'sdisease). 5. Enrolment in another clinical trial with use of experimental therapeutic agents.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female subjects scheduled to undergo left heart catheterization or peripheral angiography at LSUHSC Shreveport cardiac catheterization laboratory will be given the opportunity to participate. Controls will be recruited via flyers posted in various parts of LSUHSC Shreveport.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2013-09; Primary Completion 2017-05-07 (Actual); Study Completion 2017-05-07 (Actual)

PRIMARY OUTCOMES:
Free Sulfide, Bound Sulfide and Acid Labile Sulfide | 1 year
  Unit of Measure: nMol

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kevil, PhD, Principal Investigator — LSUHSC Shreveport
Locations (1):
- LSUHSC, Shreveport, Louisiana, United States

REFERENCES:
- [Background] Mosca L, Ferris A, Fabunmi R, Robertson RM; American Heart Association. Tracking women's awareness of heart disease: an American Heart Association national study. Circulation. 2004 Feb 10;109(5):573-9. doi: 10.1161/01.CIR.0000115222.69428.C9. Epub 2004 Feb 4. PMID 14761901
- [Background] Hirsch AT, Allison MA, Gomes AS, Corriere MA, Duval S, Ershow AG, Hiatt WR, Karas RH, Lovell MB, McDermott MM, Mendes DM, Nussmeier NA, Treat-Jacobson D; American Heart Association Council on Peripheral Vascular Disease; Council on Cardiovascular Nursing; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Surgery and Anesthesia; Council on Clinical Cardiology; Council on Epidemiology and Prevention. A call to action: women and peripheral artery disease: a scientific statement from the American Heart Association. Circulation. 2012 Mar 20;125(11):1449-72. doi: 10.1161/CIR.0b013e31824c39ba. Epub 2012 Feb 15. No abstract available. PMID 22343782
- [Background] Shen X, Pattillo CB, Pardue S, Bir SC, Wang R, Kevil CG. Measurement of plasma hydrogen sulfide in vivo and in vitro. Free Radic Biol Med. 2011 May 1;50(9):1021-31. doi: 10.1016/j.freeradbiomed.2011.01.025. Epub 2011 Jan 27. PMID 21276849
- [Background] Shen X, Peter EA, Bir S, Wang R, Kevil CG. Analytical measurement of discrete hydrogen sulfide pools in biological specimens. Free Radic Biol Med. 2012 Jun 1-15;52(11-12):2276-83. doi: 10.1016/j.freeradbiomed.2012.04.007. Epub 2012 Apr 19. PMID 22561703